CLINICAL TRIAL: NCT00862147
Title: The Effect of the International Child Development Program - A Randomised Controlled Trial
Brief Title: Effectiveness Study of the International Child Development Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was stopped due to failure to recruit sufficient participants
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4.2006.2381
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Psychosocial Functioning; Child Development
Keywords: Child psychosocial Functioning
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICDP (Experimental): International Child Development Program
  Interventions: Behavioral: ICDP
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: ICDP — Parent training group
  Other Names: International Child Development Program
  Arms: ICDP
Behavioral: Treatment as usual — Parent and/or child focused interventions
  Arms: Treatment as usual

SUMMARY:
The objective of this study is to evaluate the effect of the International Child Development Program (ICDP). Research questions to be answered:

1. Does the ICDP affect children's psychosocial functioning compared to treatment as usual?
2. Does the ICDP change parent-child interaction?

ELIGIBILITY:
Inclusion Criteria:

* SDQ >/= 9, subjective treatment need

Exclusion Criteria:

* Already in treatment

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
psychosocial functioning | study terminated

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wichstrom, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway